CLINICAL TRIAL: NCT00479297
Title: Ascending Single Dose Study of the Safety, Tolerability, Pharmacokinetics (PK), and Pharmacodynamics (PD) of SAM-531 Administered Orally to Healthy Japanese Male Subjects
Brief Title: Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SAM-531 in Healthy Japanese Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3193A1-101
Record Dates: First submitted 2007-05-24; First posted 2007-05-28 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — SAM-531

INTERVENTIONS:
Drug: SAM-531

SUMMARY:
To assess the safety and tolerability of ascending single oral doses of SAM-531, an investigational drug, in healthy Japanese male subjects. Secondary: To obtain preliminary pharmacokinetic (PK) and pharmacodynamic (PD) profiles of SAM-531 in healthy Japanese male subjects.

ELIGIBILITY:
Inclusion criteria:

* Men aged 20 to 45 years (inclusive) at the time of getting informed consent.
* Body mass index (BMI) in the range of 17.6 to 26.4 kg/m2 and body weight ≥50 kg (BMI = [weight (kg)]/[height (m)2).
* Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and digital 12-lead electrocardiogram (ECG). Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and creatinine levels must be within the upper limit of normal for eligibility.

Exclusion criteria

* Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
* Any clinically important deviation from normal limits in physical examination, vital signs, digital 12-lead ECGs, or clinical laboratory test results.
* Consumption of any caffeine-containing products (e.g., coffee, tea, chocolate, or soda) or alcoholic beverages is prohibited from 48 hours and consumption of grapefruit or a grapefruit-containing product is prohibited from 72 hours before study day 1.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72
Dates: Start 2006-05; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability

SECONDARY OUTCOMES:
Pharmacokinetics and pharmacodynamics

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer